CLINICAL TRIAL: NCT07105722
Title: A Phase 1, Observer-Blind, Randomized, Active Controlled Trial to Evaluate the Safety and Immunogenicity of An Investigational Pneumococcal Vaccine in Adults 50 To 64 Years of Age
Brief Title: A Trial to Evaluate the Safety and Immune Response of an Investigational Pneumococcal Vaccine in Adults 50 To 64 Years of Age
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 221544
Record Dates: First submitted 2025-08-04; First posted 2025-08-06 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Pneumonia, Bacterial
Keywords: Streptococcus pneumoniae; Pn-MAPS30plus; 20 valent pneumococcal conjugate vaccine (PCV20)
MeSH Terms: conditions — Pneumonia, Bacterial

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This trial will be conducted in an observer-blind manner.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pn-MAPS30plus Group (Experimental): Participants receive a single dose of Pn-MAPS30plus on Day 1.
  Interventions: Biological: Pn-MAPS30plus
- PCV20 Group (Active Comparator): Participants receive a single dose of PCV20 on Day 1.
  Interventions: Combination Product: PCV20

INTERVENTIONS:
Biological: Pn-MAPS30plus — The Pn-MAPS30plus vaccine will be administered intramuscularly.
  Arms: Pn-MAPS30plus Group
Combination Product: PCV20 — The PCV20 vaccine will be administered intramuscularly.
  Arms: PCV20 Group

SUMMARY:
This clinical study is designed to evaluate an investigational pneumococcal vaccine named Pn-MAPS30plus. The vaccine is designed to stimulate the immune system to produce antibodies against various serotypes of the S. pneumoniae bacteria, potentially aiding the body in fighting infection upon exposure. Pn-MAPS30plus aims to broaden protection by covering more serotypes than currently licensed pneumococcal vaccines. The study's purpose is to determine whether the vaccine is safe, well-tolerated, and effective in inducing immune responses against S. pneumoniae.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
2. Written or witnessed/thumb printed informed consent obtained from the participant prior to performance of any trial-specific procedure.
3. Healthy male and female participants between and including 50 through 64 YOA at the time of Informed consent form (ICF) signature.
4. Female participants of childbearing potential may be enrolled if they practice adequate contraception and have a negative pregnancy test prior to study intervention administration.

Exclusion Criteria:

1. History of microbiologically proven Invasive Pneumococcal Disease (IPD) caused by S. pneumoniae within the past 3 years.
2. History of any reaction or hypersensitivity likely to be exacerbated by any component of the study intervention(s).
3. Any confirmed or suspected immunosuppressive or immunodeficient condition.
4. Hypersensitivity to latex.
5. Clinical conditions representing a contraindication to intramuscular vaccination, and blood collection.
6. Documented history of Human immunodeficiency virus (HIV)-positive participant.
7. Acute or unstable chronic clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, or metabolic conditions as determined by the investigator.
8. Recurrent history of uncontrolled neurological or any neuroinflammatory disorders.
9. Any behavioural or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with trial participation.
10. History of potential immune-mediated disorders (pIMDs).
11. Any other clinical condition that, might pose additional risk to the participant.
12. Use of any investigational or non-registered product other than the study interventions during the period beginning 30 days before the study intervention administration.
13. History of previous vaccination with any pneumococcal vaccine.
14. Receipt of blood or plasma products or immunoglobulins, from 90 days before study intervention administration, or planned receipt within 30 days of study intervention administration.
15. Chronic administration of immune-modifying drugs (defined as more than 14 consecutive days in total) and/or planned use of long-acting immune-modifying treatments at any time up to the end of the trial.
16. Pregnant or lactating female participant.
17. History of chronic alcohol consumption and/or drug abuse, based on investigator judgment.

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 127 (Actual)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-06-09 (Estimated); Study Completion 2026-06-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Each Solicited Administration Site (Local) Event | Day 1 (post-vaccination) to Day 7
Number of Participants with Each Solicited Systemic Event | Day 1 (post-vaccination) to Day 7
Number of Participants with Any Unsolicited Adverse Events (AEs) | Day 1 (post-vaccination) to Day 30
Number of Participants with Serious AEs (SAEs), Adverse Events of Special Interest (AESIs) and AEs Leading to Withdrawal | Day 1 up to trial end (Month 6)
Number of Participants with Hematological and Biochemical Laboratory Abnormalities | On Day 8

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - GSK Investigational Site, Norwood, South Australia
  - GSK Investigational Site, Bayswater, Victoria
  - GSK Investigational Site, Camberwell, Victoria
  - GSK Investigational Site, East Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf